CLINICAL TRIAL: NCT03483935
Title: Microwave Therapy for Treatment of Precancerous Actinic Keratoses
Acronym: MTAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Emblation Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016DS12
Record Dates: First submitted 2018-02-22; First posted 2018-03-30 (Actual); Results first posted 2021-02-23 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2022-05

CONDITIONS: Actinic Keratoses; Precancerous Skin Lesion
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Intervention Model Description: Randomised, internally controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microwave energy treatment (Experimental): The microwave treatment will be delivered using the microwave instrument, SWIFT, manufactured by Emblation and CE marked for this indication, will be used to deliver the microwave treatment. The microwave dose will be between 2 Watt and 4 Watt. The treatment will consist of 3, 2 to 3 second bursts delivered to the same lesion with 5-20 seconds between bursts.
  Interventions: Other: Microwave treatment
- Control (No Intervention): No treatment will be given.

INTERVENTIONS:
Other: Microwave treatment — Microwave energy delivered using the microwave instrument, SWIFT, manufactured by Emblation and CE marked for dermatology applications.
  Arms: Microwave energy treatment

SUMMARY:
This is a two-stage feasibility study to determine if focussed microwave energy is a suitable treatment for Actinic Keratoses (AK).

The two study stages are as follows:

Stage 1:

To determine the electrical properties of permittivity in AK on the hand and bald scalp for subsequent optimisation of the SWIFT instrument to provide the correct dose of microwave energy to the AK.

Stage 2:

1. Evaluate the efficacy of microwave energy as a treatment for AK
2. Evaluate the long-term resolution of AK following microwave treatment
3. Assess the feasibility and acceptability of using microwave energy as a treatment for AK
4. Identify the potential mode of action of microwave energy in the treatment of AK.

The primary objective is to evaluate the efficacy of microwave therapy versus no treatment on the resolution of AK lesions using visual assessment. The primary outcome measure is full or partial resolution of the AK assessed by skin examination.

DETAILED DESCRIPTION:
This study is a collaboration between the University of Dundee, NHS Tayside and Emblation Ltd, funded by Innovate UK. Emblation is a Scottish based Small Medium sized Enterprise (SME) and is an established global leader in the design, development and manufacture of microwave medical devices.

Actinic keratoses (AK) are believed the most common pre-cancerous lesions in humans and are precursors to invasive cutaneous squamous cell carcinoma (cSCC), a malignancy that has more than doubled in incidence in the UK in the last decade due to ageing populations and increased UV exposure (Goon 2017). The UK incidence of cSCC now exceeds 30,000 annually (estimated >50,000 cases/year, Public Health England, unpublished data) with significant health burden and NHS costs These skin cancers are often multiple, especially in immunosuppressed high-risk populations. AK are very common "sun damage" skin lesions found on sun-exposed areas of the skin, such as the backs of hands and bald scalp. Up to 70% of our elderly population have AK and 65% of cSCC arise from previously identified AK. AK are readily identified clinically so AK treatment offers an important opportunity for cancer prevention, but our ability to treat is limited by undesirable local adverse reactions from existing topical treatments which fail to balance effectiveness, side effects and cost. None of the currently available treatments for AK are suitable for widespread use in the community and are only partially effective. Other more effective treatments such as photodynamic therapy are expensive and time consuming and need to be delivered by experts in secondary care. NHS dermatologists are already overburdened and elderly patients with AK do not wish to travel. AK therapy would be greatly improved by a cheap, convenient, well-tolerated and efficacious therapy that can be delivered closer to home by General Practitioners (GPs) or nurses.

Clinically, AK display a spectrum of severity from mild Grade 1 lesions, which are just visible and just (barely) palpable, through Grade 2 red and scaly lesions (easily felt and seen), to the most severe Grade 3 lesions, which are grossly hyperkeratotic and "thickened" skin lesions. In practice, it is easier to grade them as 'thin' (just palpable) or 'thick' (with substance to them). It is possible that the dielectric properties of Thick and Thin AK will differ and therefore the measurement study will need to be carried out on both types of AK such that the appropriate microwave dose can be given to these variable skin lesions

The investigator's hypothesis is that localised microwave energy therapy is a suitable treatment for Actinic Keratosis (AK) skin lesions.

The use of microwave technology is well established as ablative doses for treatment of malignancy e.g. hepatocellular carcinoma. There are no known studies using microwave for treatment of pre-cancerous skin conditions or skin cancers. Furthermore, there is very little understanding of the biological process evoked by localised microwave exposure in the skin or of the clinically-relevant biological mechanisms triggered.

Emblation already have a CE-marked microwave instrument used successfully for the treatment of plantar viral warts, the SWIFT device. The investigators now wish to undertake a feasibility trial in 12 participants, each with multiple AK on dorsal hand skin or bald scalp or both. The trial will examine the tolerability, acceptability, efficacy and long-term resolution of AK following one or more treatments with microwave energy delivered using the SWIFT device.

Previous studies performed by Emblation using SWIFT on plantar viral warts found it to be effective and safe. Some participants experienced minor discomfort during the microwave therapy but any pain stopped when treatment stopped. Some reddening of the skin at the treatment site may occur but this resolved after 24 hours. Some instances of a haematoma have been seen at larger doses, typically resolving within 7 days.

This will be a two-stage study, stage 1 to measure the electrical properties of AKs in patients. The data from stage 1 allows derivation of the power settings to be used with SWIFT for AK in stage 2, to conduct a randomised controlled trial of microwave treatment, delivered using SWIFT, versus no treatment.

The SWIFT device has variable power and duration controls, the protocol suitable for plantar viral warts is unlikely to be compatible with AK. Plantar warts (verrucas) are considerably thicker than AK and are located on much thicker, more robust areas of normal skin. AK are most common in the elderly population and are located on thinner, more delicate skin. The investigators therefore anticipate that AK will require a smaller dose of microwave energy than plantar warts. In order to derive the correct power and duration settings for the Swift instrument and impart the correct amount of electromagnetic energy (referred to as dose) into the AK, the dielectric properties of AK need to be determined to confirm how the specific tissue responds to the electromagnetic energy (microwave). By measuring relative permittivity (commonly abbreviated to Epsilon relative Er) the dielectric properties of the AK can be determined.

The established method of measurement requires the tissue/material under test to come into contact with a specially designed probe attached to an instrument that measures the response to a radiated signal at the same frequency (8GHz) as that used in Emblation's product "Swift". There are a number of instrument and probe manufacturers e.g. Keysight (HP/Agilent), SPEAG, Anritsu. The probe can be used to test solids, liquids and biological tissues by placing the probe in direct contact for a few seconds whilst remaining still during data acquisition by the instrument.

The instrument (Anritsu MS46122A) providing the probe excitation conforms to the following standards: CE Mark, Low voltage (2006/95/EC) and Safety (EN 61010-1:2010). The energy imparted into the lesion for the measurement will not exceed 0.5mW, by way of comparison this is far less than a mobile phone (up to 500mW) and a FitBit (1.6mW) thus there is no inherent danger to the volunteer.

Emblation employees will operate the instruments and direct the subjects to the probe. Other study team staff may work in conjunction with NHS staff at the time of recruitment and/or at the time of measurement.

Microwave energy is converted to heat in the skin layers and forms the basis of the therapy. The target temperature of 43-46 degrees Centigrade is crucial in eliciting the correct immune response in the tissue. As the current instrument is 'tuned' with an antenna for plantar warts, it may not be as efficient at imparting the energy into the AK lesions and the target temperature may not be achieved with the same power and duration settings. Conversely, if the AK provides a more efficient conversion of microwave to temperature, potentially too high a temperature may be reached at a given power and duration combination. Stage 1 data will be analysed to model the efficiency of the current antenna in computer simulations and values for input power (W) and duration (s) will be derived from the modelling data, subsequently to be used in the stage 2 of the trial. This will provide the correct dose of microwave energy to be used in Stage 2.

Once the settings required for AK have been determined, participants will be recruited into Stage 2 in order to determine efficacy, long term resolution, tolerability and potential mode of action of microwave treatment for AK.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants
* Age 18 years and over
* Clinical diagnosis of precancerous Actinic Keratosis made by a dermatologist
* Able to perform study assessments

Exclusion Criteria:

* Inability to give informed consent
* Implantable Cardioverter-defibrillator (ICD), pacemaker or other implantable device
* Metal implants at site of treatment
* Known allergy or intolerance to microwave therapy
* Unstable co-morbidities (cardiovascular disease, active malignancy, vasculopathy, inflammatory arthritis) which, in the opinion of the Chief Investigator (CI), would make the patient unsuitable to be enrolled in the study.
* Individuals who are immunosuppressed (organ transplant recipients, haematologic malignancies, HIV).
* Individuals will not be enrolled to the study if they are participating in the clinical phase of another interventional trial or have done so within the last 30 days. Individuals who are participating in the follow-up phase of another interventional trial, or who are enrolled in an observational study, will be co-enrolled where the CIs of each study agree that it is appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Proby, MBCHB, Principal Investigator — University of Dundee
Locations (1):
- NHS Tayside, Dundee, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bristow I, Lim WC, Lee A, Holbrook D, Savelyeva N, Thomson P, Webb C, Polak M, Ardern-Jones MR. Microwave therapy for cutaneous human papilloma virus infection. Eur J Dermatol. 2017 Oct 1;27(5):511-518. doi: 10.1684/ejd.2017.3086. PMID 29084638
- [Background] Criscione VD, Weinstock MA, Naylor MF, Luque C, Eide MJ, Bingham SF; Department of Veteran Affairs Topical Tretinoin Chemoprevention Trial Group. Actinic keratoses: Natural history and risk of malignant transformation in the Veterans Affairs Topical Tretinoin Chemoprevention Trial. Cancer. 2009 Jun 1;115(11):2523-30. doi: 10.1002/cncr.24284. PMID 19382202
- [Background] Eder J, Prillinger K, Korn A, Geroldinger A, Trautinger F. Prevalence of actinic keratosis among dermatology outpatients in Austria. Br J Dermatol. 2014 Dec;171(6):1415-21. doi: 10.1111/bjd.13132. Epub 2014 Nov 19. PMID 24864059
- [Background] Goon PK, Greenberg DC, Igali L, Levell NJ. Squamous Cell Carcinoma of the Skin has More Than Doubled Over the Last Decade in the UK. Acta Derm Venereol. 2016 Aug 23;96(6):820-1. doi: 10.2340/00015555-2310. No abstract available. PMID 26631391
- [Background] Liang P, Wang Y. Microwave ablation of hepatocellular carcinoma. Oncology. 2007;72 Suppl 1:124-31. doi: 10.1159/000111718. Epub 2007 Dec 13. PMID 18087193
- [Background] Marks R, Rennie G, Selwood TS. Malignant transformation of solar keratoses to squamous cell carcinoma. Lancet. 1988 Apr 9;1(8589):795-7. doi: 10.1016/s0140-6736(88)91658-3. PMID 2895318
- [Background] Martin R.C.G. (2011) Microwave Ablation and Hepatocellular Carcinoma. In: McMasters K. (eds) Hepatocellular Carcinoma:. Springer, New York, NY
- [Background] Poggi G, Tosoratti N, Montagna B, Picchi C. Microwave ablation of hepatocellular carcinoma. World J Hepatol. 2015 Nov 8;7(25):2578-89. doi: 10.4254/wjh.v7.i25.2578. PMID 26557950
- [Background] Wang T, Lu XJ, Chi JC, Ding M, Zhang Y, Tang XY, Li P, Zhang L, Zhang XY, Zhai B. Microwave ablation of hepatocellular carcinoma as first-line treatment: long term outcomes and prognostic factors in 221 patients. Sci Rep. 2016 Sep 13;6:32728. doi: 10.1038/srep32728. PMID 27620527

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited to the Stage 1, dose finding study in March 2018.
  Participants were recruited to Stage 2, the RCT, between May 2018 and October 2018.
  Participants for both stages were recruited from the Department of Dermatology, Ninewells Hospital, NHS Tayside, UK.
Units Other Than Participants: Number of AK Lesions
Groups:
- Trial Population: Stage 1: Determine the electrical properties of AKs Stage 2: Evaluate the efficacy of microwave energy as a treatment for AK
Period: Stage 1: Dose Setting Study
Arm/Group | Trial Population
Started | 7; 34 Number of AK Lesions
Completed (7 participants were recruited to the stage 1, dose finding study) | 7; 34 Number of AK Lesions
Not Completed | 0; 0 Number of AK Lesions
Period: Stage 2: Randomised Controlled Trial
Arm/Group | Trial Population
Started (Eleven participants were recruited and randomized to Stage 2. 179 AKs (93 treated, 86 untreated) were assessed.) | 11; 179 Number of AK Lesions (Participants were randomised to receiving treatment on the left or right side.)
AKs Treated | 11; 93 Number of AK Lesions
AKs Not Treated | 11; 86 Number of AK Lesions
Completed | 11; 179 Number of AK Lesions
Not Completed | 0; 0 Number of AK Lesions

BASELINE CHARACTERISTICS:
Population: History of skin cancer was not collected for Dose Finding population History of other cancer was not collected for the Dose Finding population
Groups:
- Dose Finding Population: Consented participants had the electric properties of permittivity in AK on hand and bald scalp assessed for subsequent optimisation of the dose of microwave therapy to be used in the RCT.
- RCT Study Population: This was a randomized, internally controlled, feasibility study. Consented participants had the treatment site (scalp/forehead or hands) selected based on a clinical decision. Participants were randomized to treatment to the left or right side.
  The microwave treatment was delivered using the microwave instrument, SWIFT, manufactured by Emblation and CE marked for this indication. The microwave dose was between 2 Watt and 4 Watt. The treatment will consist of 3, 2 to 3 second bursts delivered to the same lesion with 5-20 seconds between bursts.
  No treatment was administered to the control side.
- Total: Total of all reporting groups
Arm/Group | Dose Finding Population | RCT Study Population | Total
Number analyzed (Participants) | 7 | 11 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (7) | 78 (6) | NA (NA) — Different patient populations for stage 1 and stage 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 5 | 7 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
History of skin cancer [Count of Participants; unit: Participants] — Population: Data were not collected
  Participants
    number analyzed (Participants) | 0 | 11 | 11
    (all) | 0 | 10 | 10
History of other cancer [Count of Participants; unit: Participants] — Population: Data were not collected
  Participants
    number analyzed (Participants) | 0 | 11 | 11
    (all) | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Resolution of AK Lesions Following Microwave Treatment
Description: The resolution of each treated AK lesion will be determined by clinical assessment. Resolution is predetermined as either partial (resolution of the area covered by the microwave probe, but with a rim or persistent AK) or full (complete resolution of the entire AK) over all time periods. Response will be assessed at visits 3 (day 8), 4 (day 15), 6 (day 28), 8 (day 42), 10 (day 60) and 11 (day 120). Mixed-effects logistic regression models analysed the effect of microwave therapy with random effects for participant and visit (≤ 6 per participant). Each visit will be analysed as a categorical variable as they were spaced unequally in time. Variables representing sex, age, skin site (hand/scalp) and AK subtype (thick/thin) will be included as covariates. The data reported in the outcome table is the number of resolved AK lesions.
Time Frame: Baseline, day 8, 15, 28, 42, 60 and 120
Population: Eleven participants were randomized and 179 AKs (93 treated, 86 untreated) assessed. All participants completed treatment as planned.
Measure: Count of Units; unit: AK lesions
Units Other Than Participants: AK lesions
Groups:
- Microwave Energy Treatment: Microwave dose for participants 1 and 2 was 5 Watt. Dose for participants 3 through 9 was between 2 Watt and 4 Watt. Treatment consists of 3, 2 to 3 second bursts of microwave energy, delivered to the same lesion with 5-20 seconds between bursts.
- Control: No treatment
Arm/Group | Microwave Energy Treatment | Control
Number analyzed (Participants) | 11 | 11
Number analyzed (AK lesions) | 93 | 86
AK lesions
  Day 8 | 73 | 2
  Day 15 | 73 | 7
  Day 28 | 86 | 9
  Day 42 | 86 | 9
  Day 60 | 81 | 11
  Day 120 | 84 | 13

2. Primary Outcome: Complete Resolution of AKs Following Microwave Treatment
Description: The resolution of each treated AK lesion will be determined by clinical assessment. Resolution is predetermined as either partial (resolution of the area covered by the microwave probe, but with a rim or persistent AK) or full (complete resolution of the entire AK) over all time periods. Treatment will be given at day 1, with a second treatment on day 28 based on a clinical decision. Response will be assessed at visits 3 (day 8), 4 (day 15), 6 (day 28), 8 (day 42), 10 (day 60) and 11 (day 120). Clinical photos will be taken at each hospital visit. Mixed-effects logistic regression models analysed the effect of microwave therapy with random effects for participant and visit (≤ 6 per participant). Each visit will be analysed as a categorical variable as they were spaced unequally in time. Variables representing sex, age, skin site (hand/scalp) and AK subtype (thick/thin) will be included as covariates.
Time Frame: Baseline, day 8, 15, 28, 42, 60 and 120
Population: as for outcome 1
Measure: Count of Units; unit: Number of lesions
Units Other Than Participants: Number of lesions
Arm/Group | Microwave Energy Treatment | Control
Number analyzed (Participants) | 11 | 11
Number analyzed (Number of lesions) | 93 | 86
Number of lesions
  Day 8 | 4 | 1
  Day 15 | 7 | 1
  Day 28 | 20 | 2
  Day 42 | 23 | 3
  Day 60 | 41 | 5
  Day 120 | 39 | 6

3. Primary Outcome: Partial Resolution of AKs Following Microwave Treatment
Description: as for outcome 2
Time Frame: Baseline, day 8, 15, 28, 42, 60 and 120
Population: as for outcome 1
Measure: Count of Units; unit: Number of Lesions
Units Other Than Participants: Number of Lesions
Arm/Group | Microwave Energy Treatment | Control
Number analyzed (Participants) | 11 | 11
Number analyzed (Number of Lesions) | 93 | 86
Number of Lesions
  Day 8 | 69 | 1
  Day 15 | 66 | 6
  Day 28 | 66 | 7
  Day 42 | 63 | 6
  Day 60 | 40 | 6
  Day 120 | 45 | 7

4. Secondary Outcome: Level of Pain Experienced During Treatment
Description: To evaluate the safety and tolerability of microwave treatment as a therapy for AK, participants were asked about level of pain during treatment. Participants were asked to rate their pain level during each treatment as i) mild, ii) moderate or iii) severe.
Time Frame: Treatment 1 (day 1) and treatment 2 (day 28)
Population: 11 participants had a total of 93 AKs treated at visit 1 (day 1), with 10 participants having a total of 51 of the original 93 AKs receiving a second treatment at visit 6 (day 28).
Measure: Number; unit: Number of AK lesions treated
Units Other Than Participants: Number of AK lesions treated
Groups:
- Treatment 1: First microwave treatment, administered at visit 1, day 1
- Treatment 2: Second microwave treatment, administered at visit 6, day 28
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 11 | 10
Number analyzed (Number of AK lesions treated) | 93 | 51
Number of AK lesions treated
  Mild pain during treatment | 7 | 5
  Moderate pain during treatment | 32 | 27
  Severe pain during treatment | 54 | 19

5. Secondary Outcome: Duration of Pain Post Treatment
Description: To evaluate the safety and tolerability of microwave treatment as a therapy for AK, participants were asked about the duration of pain immediately after each treatment. Duration was grouped into 5 pre-determined periods, i) few seconds, ii) up to 5 minutes, iii) up to 10 minutes, iv) up to 20 minutes and v) over 30 minutes. The decision to administer a second treatment was made by the investigator.
Time Frame: Treatment 1 (day 1) and Treatment 2 (day 28)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 11 | 10
Participants
  Duration: Few seconds | 7 | 8
  Duration: Up to 5 minutes | 2 | 2
  Duration: Up to 10 minutes | 1 | 0
  Duration: Up to 20 minutes | 1 | 0
  Duration: Over 30 minutes | 0 | 0

6. Secondary Outcome: Change in Ki67 Staining Determined Immunohistochemically by the Use of Specific Antibodies on Fixed Material
Description: To identify the mode of action of microwave treatment on biomarkers of cell proliferation as a therapy for AK. Results are provided on the staining positivity scale of +, ++ and +++. The minimum value is + , meaning the least staining. The maximum value is +++, meaning the most staining identified.
Time Frame: Day 15
Population: One AK lesion from the microwave treatment allocation was pre-selected for biopsy. Biopsy taken from all participants 15 days post microwave energy treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Microwave Energy Treatment: Biopsy taken from all participants 15 days post microwave energy treatment
Arm/Group | Microwave Energy Treatment
Number analyzed (Participants) | 11
Participants
  + stain positivity | 9
  ++ stain positivity | 1
  +++ stain positivity | 1

7. Secondary Outcome: Change in Hematoxylin and Eosin Stain
Description: To identify the mode of action of microwave treatment on biomarkers of cell survival.
Time Frame: Day 15 OR day 42
Population: all participants treated with microwave therapy.
Measure: Count of Participants; unit: Participants
Groups:
- Change in Hematoxylin and Eosin Stain: all participants treated with microwave therapy.
Arm/Group | Change in Hematoxylin and Eosin Stain
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the date of consent until the participant's last study visit. For Stage 1, study duration was 1 day. For stage 2, RCT, maximum participant duration on the trial was 35 days washout period (if required) and 120 days trial duration. SAEs were followed up for both stages until 30 days after the participant's last visit.
Description: Participants were asked at every visit about the occurrence of adverse events at the site of treatment and biopsy and details of hospitalization. Expected adverse events following microwave therapy include stinging, redness, tingling, numbness or soreness. Participants were asked to score their pain immediately following microwave treatment and 30 minutes after treatment.
Groups:
- Stage 1 Dose Finding Study: To determine the electrical properties of permitivity in AK on the hand and scalp.
- Stage 2 RCT: The microwave treatment delivered using the microwave instrument, SWIFT, manufactured by Emblation and CE marked for this indication. The microwave dose was between 5 Watt for the first two participants and 2 Watt and 4 Watt for the remaining nine participants. The treatment will consist of 3, 2 to 3 second bursts delivered to the same lesion with 5-20 seconds between bursts.
Arm/Group | Stage 1 Dose Finding Study | Stage 2 RCT
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/11
Other Adverse Events (participants affected / at risk) | 0/7 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Dose Finding Study (N=7) | Stage 2 RCT (N=11)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Fracture of distal tibia resulting in hospitalisation. Unrelated to intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stage 1 Dose Finding Study (N=7) | Stage 2 RCT (N=11)
Treatment administration site pain (General disorders) | 0 (0) | 11 (21) — Transient pain at site of microwave treatment administration
Treatment administration site pruritus (General disorders) | 0 (0) | 4 (6) — Transient pruritus at site of microwave treatment administration
Treatment administration site erythema (General disorders) | 0 (0) | 5 (6) — Transient erythema at site of microwave treatment administration
Treatment administration site scab (General disorders) | 0 (0) | 9 (10) — Transient scabbing at site of microwave treatment administration
Treatment administration site erosion (General disorders) | 0 (0) | 2 (3) — Transient erosion at site of treatment administration
Treatment administration site exfoliation (General disorders) | 0 (0) | 3 (3) — Transient exfoliation at site of microwave treatment administration
Skin tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Transient skin tightness at site of microwave treatment administration
Treatment administration site paraesthesia (General disorders) | 0 (0) | 1 (1) — Transient paraesthesia at microwave treatment site
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Transient headache post microwave treatment
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Injury to scab at site of treatment administration unrelated to intervention
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) — Unrelated to intervention
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) — Unrelated to intervention
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) — Unrelated to intervention
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) — Unrelated to intervention
Paronychia (Infections and infestations) | 0 (0) | 1 (1) — Unrelated to intervention
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to intervention
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Unrelated to intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT03483935/Prot_001.pdf
  • Statistical Analysis Plan (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT03483935/SAP_002.pdf